CLINICAL TRIAL: NCT05934331
Title: An Open-label, Multicenter Phase II Clinical Study to Evaluate the Efficacy, Safety, and Tolerability of the LM-302 Combination With Other Anti-tumor Treatment in Subjects With CLDN18.2-positive Advanced Gastro-Intestinal Cancer.
Brief Title: A LM-302 Combination With Other Anti-Tumor Therapies Phase ll Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Zhejiang Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: LaNova Medicines Limited (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM302-02-201
Record Dates: First submitted 2023-06-19; First posted 2023-07-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Malignant Neoplasms of Digestive Organs
MeSH Terms: interventions — toripalimab; Capecitabine; Tegafur; gimeracil; potassium oxonate; Nivolumab; apatinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LM-302 in combination with Toripalimab (Experimental)
  Interventions: Drug: LM-302; Drug: Toripalimab
- LM-302 in combination with other therapies (Experimental)
  Interventions: Drug: LM-302; Drug: Toripalimab; Drug: Capecitabine; Drug: Tegafur, Gimeracil and Oteracil Potassium Capsules; Drug: Nivolumab; Drug: Apatinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: LM-302 — Q2W/Q3W，Administered intravenously
Drug: Toripalimab — Q2W/Q3W,Administered intravenously
Drug: Capecitabine — BID,Oral Administration
  Arms: LM-302 in combination with other therapies
Drug: Tegafur, Gimeracil and Oteracil Potassium Capsules — BID,Oral Administration
  Arms: LM-302 in combination with other therapies
Drug: Nivolumab — Q4W,Administered intravenously
  Arms: LM-302 in combination with other therapies
Drug: Apatinib — QD,Oral Administration
  Arms: LM-302 in combination with other therapies
Drug: Gemcitabine — Q4W,Administered intravenously
  Arms: LM-302 in combination with other therapies

SUMMARY:
This study is to evaluate the efficacy of the LM-302 Combination With Other Therapies in patients with CLDN18.2-positive Advanced Digestive Tract Tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Aged 18-80 years old (including boundary values) .
3. Eastern Cooperative Oncology Group (ECOG) performance status of0-1.
4. Life expectancy ≥ 3 months.
5. Subjects with advanced gastrointestinal tumors diagnosed histologically and/or cytologically and who have failed or are intolerant to prior standard first-line therapy (imaging confirmation required)
6. CLDN18.2-positive subjects.
7. At least one measurable lesion.
8. Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose.
9. Subjects who are able to communicate well with investigators and understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Subjects with known HER2-positive gastric cancer/adenocarcinoma of the gastroesophageal junction
2. Subjects have participated in any other clinical trial within 28 days prior to 1st dosing of investigational medicinal product (IMP).
3. Subjects with anti-tumor treatment within 21 days prior to 1st dosing of IMP.
4. Previous immunotherapy and grade ≥3 irAE or grade ≥2 immune-related myocarditis. (for cohorts treated with combination PD-1).
5. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
6. Present peripheral sensory or motor neuropathy ≥ grade 2.
7. Subjects with uncontrolled pain.
8. Subjects with symptomatic/active central nervous system(CNS)metastases.
9. Subject who have uncontrollable third space effusion.
10. Subjects with known hypersensitivity to antibody therapy.
11. Subjects have treated with the same target.
12. Subjects have received Strong inhibitor/strong inducer of CYP3A4 within 14 days prior to first dose.
13. Use of any live vaccines within 28 days prior to 1st dosing of IMP.
14. Subjects with current or previous interstitial lung diseases or pneumonia requiring oral or intravenous glucocorticoids for adjuvant therapy.
15. Subjects on anticoagulants, such as heparin and vitamin K antagonists.
16. Clinically uncontrollable persistent recurrent vomiting.
17. Uncontrollable/severe gastrointestinal bleeding, ulceration or diarrhea within 28 days prior to first dose of IMP.
18. Subjects who received major surgery or interventional treatment within28 days prior to the first dosing of IMP.
19. Subjects who have other cancers, other than the one treated in this trial, within 2 years prior to screening.
20. Subjects who have severe cardiovascular disease.
21. Subjects who have uncontrolled or severe illness.
22. Subjects who take systemic corticosteroids (> 10 mg daily prednisone equivalents) or other systemic immunosuppressive medications within 2 weeks prior to the first dosing of IMP.
23. Subjects with a known history of autoimmune diseases.
24. Subjects who have a history of immunodeficiency disease.
25. Subjects with HIV infection, active HBV or HCV infection.
26. Child-bearing potential female who have positive results in pregnancy test within 7 days before the first dose or are lactating.
27. Subject who have a known psychiatric diseases or disorders that may affect compliance with the trial.
28. Subject who is judged as not eligible to participate in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 112 weeks
  Progression free survival according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1)

SECONDARY OUTCOMES:
ORR | 112 weeks
  Objective response rate (ORR)
DOR | 112 weeks
  Duration of response (DOR)
DCR | 112 weeks
  Disease control rate (DCR = CR + PR + SD)
OS | 112 weeks
  Overall survival (OS)
AEs | 112 weeks
  Incidence of adverse events
SAEs | 112 weeks
  Incidence of serious adverse events
Temperatures | 112 weeks
  Temperatures
Pulse in BPM | 112 weeks
  Beat per Minute
Blood Pressure | 112 weeks
  Blood Pressure in mmHg
Weight | 112 weeks
  Weight in Kg
Height | 112 weeks
  Height in centimeter
Blood Routine examination | 112 weeks
  Laboratory tests-Blood Routine examination
Urine Routine test | 112 weeks
  Laboratory tests-Urine Routine test
Blood biochemistry | 112 weeks
  Laboratory tests-Blood biochemistry
Coagulation function | 112 weeks
  Laboratory tests- Coagulation function
LVEF | 112 weeks
  Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage
HR | 112 weeks
  12-lead electrocardiogram (ECG) in HR
RR | 112 weeks
  12-lead electrocardiogram (ECG) in RR
PR | 112 weeks
  12-lead electrocardiogram (ECG) in PR
QRS | 112 weeks
  12-lead electrocardiogram (ECG) in QRS
QT | 112 weeks
  12-lead electrocardiogram (ECG) in QT
QTcF | 112 weeks
  12-lead electrocardiogram (ECG) in QTcF
ECOG score | 112 weeks
  Eastern Cooperative Oncology Group score
PK Parameter:Cmax | 112 weeks
  Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax)
PK Parameter：Tmax | 112 weeks
  PK Parameter:Time of Maximum Observed Concentration (Tmax)
PK Parameter: AUC | 112 weeks
  PK Parameter: Area Under the Concentration-time Curve(AUC)
PK Parameter: Cmax,ss | 112 weeks
  PK Parameter: Steady State Maximum Concentration(Cmax,ss)
PK Parameter: Cmin,ss | 112 weeks
  PK Parameter: Steady State Minimum Concentration(Cmin,ss)
PK Parameter: CLss | 112 weeks
  PK Parameter: Systemic Clearance at Steady State (CLss)
PK Parameter:Rac | 112 weeks
  PK Parameter: Accumulation Ratio (Rac)
PK Parameter: t1/2 | 112 weeks
  PK Parameter: Elimination Half-life (t1/2)
PK Parameter: Vss | 112 weeks
  PK Parameter: Volume of Distribution at Steady-State (Vss)
PK Parameter: DF | 112 weeks
  PK Parameter: Degree of Fluctuation (DF)
Immunogenicity of LM-302 | 112 weeks
  Anti-Drug antibody and Nab (if neccessary) will be tested.
Biomarker correlation | 112 weeks
  For the detection of CLDN18.2 and PD-L1
AE/SAE | 112 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai East Hospital; Jieer Ying, Principal Investigator — Zhejiang Cancer Hospital; Haiping Jiang, Principal Investigator — Zhejiang University; Rushen Zhao, Principal Investigator — Zibo Municipal Hospital; Chunmei Bai, Principal Investigator — Peking Union Medical College Hospital; Hongming Pan, Principal Investigator — Sir Run Run Shaw Hospital; Jing Dai, Principal Investigator — Zhongnan Hospital; Yiping Mou, Principal Investigator — Zhejiang Provincial People's Hospital; Haijiao Yan, Principal Investigator — The First People's Hospital of Changzhou; Aiping Zhou, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Xianglin Yuan, Principal Investigator — Tongji Hospital; Yabin Xia, Principal Investigator — First Affiliated Hospital of Wannan Medical College; Mingzhu Huang, Principal Investigator — Fudan University; Lixin Wan, Principal Investigator — Nanyang Central Hospital; Jun Zhou, Principal Investigator — Shanghai Gaobo Cancer Hospital; Youwei Zhang, Principal Investigator — Xuzhou Central Hospital; Ning Wu, Principal Investigator — Shanghai Pudong New District Gongli Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, China